CLINICAL TRIAL: NCT07113262
Title: A Multicenter, Randomized, Double-masked, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of IBI311 in Subjects With Inactive Thyroid Eye Disease
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of IBI311 in Subjects With Inactive Thyroid Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI311A302
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teprotumumab N01 injection (code name IBI311) (Experimental)
  Interventions: Drug: IBI311
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBI311 — Teprotumumab N01 injection (code name IBI311)
  Arms: Teprotumumab N01 injection (code name IBI311)
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
A multicenter clinical study to evaluate the efficacy and safety of IBI311 in subjects with inactive thyroid eye disease. The study consists of two parts, with a maximum duration of approximately 64 weeks.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-masked, placebo-controlled Phase III clinical study in inactive TED subjects. Approximately 111 eligible subjects will be randomly assigned to the IBI311 group and the placebo group in a 2:1 ratio on Day 1. The study consists of two parts, with a maximum duration of approximately 64 weeks. Part 1 includes a screening period and a double-masked treatment period, lasting for a total of approximately 28 weeks. Part 2 is a follow-up/open treatment period, lasting for up to approximately 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1.At screening and baseline, the following diagnostic criteria for inactive TED were met:

1. CAS of both eyes ≤ 2 points during the screening period and baseline;
2. According to the subject's medical history, CAS of both eyes ≤ 2 points at least 6 months before screening, or according to the subject's chief complaint or medical history, with all of the following characteristics: no progression of proptosis and no new diplopia caused by TED at least 6 months before screening or no progression of diplopia caused by TED and no new inflammatory TED symptoms;
3. According to the subject's chief complaint or medical history, the first TED diagnosis before screening was ≥ 2 years and < 10 years.

2.At baseline, the proptosis of the study eye was ≥20 mm. 3.If the subject is a female, she should be infertile or have a negative blood pregnancy test during the screening period and agree to take contraceptive measures from the screening period to 120 days after the last medication. If the subject is a male, he should agree to take contraceptive measures from the screening period to 120 days after the last medication.

Exclusion Criteria:

Subjects who meet any of the following conditions will not be eligible to participate in this study:

1. At baseline, the eyeball protrusion of the study eye decreased by ≥2 mm compared with the screening period;
2. Subjects who have been previously diagnosed with DON, or who are determined by the investigator to have DON during screening (defined as: orbital MRI/CT showing orbital apex crowding or optic nerve compression, and at least 2 of the following ophthalmological examination abnormalities that cannot be explained by other reasons: ① best corrected visual acuity [BCVA] < 0.8 or BCVA decreased by ≥ 2 lines compared with before the onset; ② abnormal pupillary light reflex or relative pupillary afferent disorder; ③ color vision abnormalities; ④ optic disc edema and optic disc pallor on fundus examination; ⑤ visual field loss; ⑥ visual evoked potential with prolonged latency and/or decreased amplitude);
3. Patients with corneal ulcers that are judged by the researchers to have no relief after treatment;
4. Planned to receive orbital radiotherapy or surgical treatment for TED (including orbital decompression, strabismus correction, eyelid correction, etc.) at any time before baseline or during the study period;
5. Poorly controlled thyroid function, defined as free triiodothyronine (FT3) or free thyroxine (FT4) deviating from the normal reference value range of the local research center laboratory by more than 50% during screening;
6. Any other diseases, metabolic disorders, abnormal physical examination or clinical laboratory test results, and there is reason to suspect that there may be diseases or conditions that may lead to contraindications to the use of the trial drug, affect the interpretation of the study results, or put the subjects at high risk of treatment complications, including but not limited to: confirmed or clinically suspected inflammatory bowel disease, coagulation disorders, history of acute cardiovascular and cerebrovascular diseases or treatment history within 180 days before screening(including but not limited to: cerebrovascular accident, transient ischemic attack, acute myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention [except diagnostic angiography], severe arrhythmia, etc.), history of malignant tumors treated or untreated in the past 5 years (except for skin squamous cell carcinoma, basal cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or thyroid papillary carcinoma that have been successfully removed and have no evidence of metastasis), severe systemic infection, proptosis not caused by TED, etc.;
7. During the screening period, any ear has: tinnitus or other history of hearing loss; or abnormal pure tone audiometry results (defined as average bone conduction hearing threshold ≥25 dB at 0.5, 1, 2, 4 kHz or bone conduction hearing threshold ≥40 dB at any frequency);
8. At screening, aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>3×ULN, or with active hepatitis B (defined as HBsAg positive with HBV-DNA load>1000 IU/mL), or receiving anti-hepatitis B virus treatment;
9. At screening, glomerular filtration rate (GFR) <30 ml/min/1.73m2 (MDRD formula: GFR = 186 × serum creatinine (mg/dl) - 1.154 × (age) - 0.203 × (0.742 [if female]), serum creatinine unit conversion: 1 μmol/L = 0.0113 mg/dL);
10. Poorly controlled diabetes at screening (defined as glycated hemoglobin ≥8.0% at screening);
11. At screening, patients have poorly controlled hypertension, with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg; renal artery stenosis; or evidence of unstable blood pressure (including orthostatic hypotension, etc.);
12. During screening, the 12-lead ECG shows a heart rate of <50 beats/min or >100 beats/min, the ECG indicates active heart disease, or the investigator believes that the ECG abnormality during screening will interfere with the interpretation of the ECG results during subsequent follow-up, especially excluding QTcF>500 ms;
13. HIV antibody or HCV antibody positive or active syphilis (defined as non-specific syphilis antibody positive or requiring anti-syphilis treatment after consultation with the infectious disease department);
14. Oral or intravenous glucocorticoids within 30 days before screening;
15. Use of glucocorticoid eye drops/eye ointment, or non-steroidal immunosuppressant eye drops within 30 days before screening;
16. Periorbital/periorbital injection of glucocorticoids within 90 days before screening;
17. Any other non-steroidal immunosuppressants taken orally or intravenously within 90 days before screening;
18. Received interleukin-6 receptor (IL-6R) antibody treatment within 180 days before screening;
19. Received CD20 antibody treatment within 1 year before screening;
20. Received IBI311 or TEPEZZA treatment at any time before screening;
21. Have received any other TED treatment drugs under development at any time before screening (including but not limited to biological agents targeting IGF-1R, FcRn, and TSHR);
22. Use of any other monoclonal antibody treatment within 90 days before screening;
23. Participated in other interventional clinical trials within 90 days before screening (for drugs, within 5 half-lives, whichever is longer; excluding vitamins and minerals), or attempted to participate in other clinical trials during the study;
24. Female subjects who are pregnant or lactating;
25. Those who are known to be allergic to the study drug ingredients, or have a history of allergies to other monoclonal antibodies; Those who are considered by the researchers to be unsuitable for participating in this clinical trial due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proptosis response rate of the study eye | 24 weeks
  Proptosis response rate (i.e., percentage of participants with a ≥ 2 mm decrease from baseline in proptosis in the study eye and without a ≥ 2 mm increase of proptosis in the fellow eye) of the study eye at Week 24

SECONDARY OUTCOMES:
Change from baseline of proptosis in the study eye | 24 weeks
  The Change from baseline of proptosis in the study eye at Week 24
Time to first achieve proptosis response in the study eye | 24 weeks
  Time to first proptosis response in the study eye at Week 24.
Change from baseline in CAS in the study eye | 24 weeks
  Change from baseline in CAS in the study eye at Week 24.
Diplopia responder rate | 24 weeks
  Diplopia responder rate (percentage of subjects with ≥ 1-grade improvement in diplopia) at Week 24.
Proptosis response rate of the fellow eye | 24 weeks
  Proptosis response rate of the fellow eye at week 24.
Change from baseline in the total score of the Graves' Ophthalmopathy Quality of Life (GO-QoL) questionnaire | 24 weeks
  Change from baseline in the total score of the Graves' Ophthalmopathy Quality of Life (GO-QoL) questionnaire at week 24.
Evaluate the safety and tolerability of IBI311 in Part 1 | up to 24 weeks
  The number, incidence, severity, and relevance to study drugs or treatments of all ocular and other systemic AEs, TEAEs, AESIs, and SAEs.
Proptosis response rate of the study eye in subjects with delayed IBI311 treatment in Part 2. | 48 weeks
  Proptosis response rate of the study eye in subjects with delayed IBI311 treatment (those who have received placebo in Part 1) in Part 2.
Proptosis response rate of the study eye in subjects with two consecutive circles of IBI311 treatment. | 48 weeks
  Proptosis response rate of the study eye in subjects with two consecutive circles of IBI311 treatment (one circle of IBI311 treatment in Part 1 and then another circle of IBI311 treatment in Part 2
Rate of disease flare/deterioration | 48 weeks
  Rate of disease flare/deterioration (The proptosis of either eye increased by ≥2 mm compared to week 24, and/or the CAS increased by ≥2 points compared to week 24 with a CAS ≥3 points) in subjects with IBI311 treatment in Part 1
Proptosis response rate of the study eye in subjects with disease flare/deterioration and receive another circle of IBI311 treatment in Part 2 | 48 weeks
  Proptosis response rate of the study eye in subjects with disease flare/deterioration after IBI311 treatment in Part 1 and then receive another circle of IBI311 treatment in Part 2.
Evaluate the safety and tolerability of IBI311 in Part 2 | through study completion, an average of 1 year
  The number, incidence, severity, and relevance to study drugs or treatments of all ocular and other systemic AEs, TEAEs, AESIs, and SAEs.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Medical University, Shenyang, Liaoning, China